CLINICAL TRIAL: NCT06874257
Title: Targeting Acute Myeloid Leukemia Immunosuppressive Microenvironment by combinedIDO1 Inhibition and PD-1 Blockade
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: TALETE-2023; 3000506 (Other Grant/Funding Number: Grant)
Record Dates: First submitted 2024-12-01; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-12

CONDITIONS: AML (Acute Myelogenous Leukemia)
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Bone Marrow, Plasm, blood, Osteo medullary biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patien with AML: The study will include untreated and newly diagnosed unfit-to-chemotherapy, adult AML patients candidate to receive the combination of venetoclax plus azacitidine according to standard clinical practice, and independently of the participation to the study. The patients will be enrolled at the time of disease diagnosis. For healthy donors, a total of 60 buffy coats will be collected in time period of 24 months. Patients who will not receive any treatment will be excluded from the study
  Interventions: Biological: Laboratory tests and in vitro studies

INTERVENTIONS:
Biological: Laboratory tests and in vitro studies — Cell models, co-culture condition set-up and functional validation, Single-cell RNA sequencing and NGS, Metabolomics analysis, metabolomics validation and intracellular metabolomics analysis, Metabolic ImmunoProfiling and epigenetic profile, CyTOF immune and signaling profiling, Monocyte, macrophages and MSCs in vitro assays.

SUMMARY:
The combination of azacitidine and venetoclax is currently considered a therapeutic strategy innovative in AML through the addition of new compounds (triplet therapies), including inhibitors of the immune checkpoint inhibitors. Despite strong motivation, the clinical results of these approaches have been disappointing overall. The mechanisms leading to treatment failure of immunotherapies in AML are poorly elucidated as the effects on the AML microenvironment induced by basic azactidine and venetoclax therapy are largely unknown. In particular, the activity of the IDO1 enzyme as a potential mechanism of microenvironment resistance has been scarcely studied. The products of the IDO1-catalysed pathway activate the signalling of the AHR in mesenchymal stem cells and enhance their immunosuppressive effects, including the ability to reprogram the phenotype of M1/M2 macrophages. Furthermore, activation of the AHR by by products of the IDO1 pathway kinurenine-promotes tolerogenic dendritic cells and the generation of regulatory T cells. Based on this rationale, TALETE-2023 will aim to analyse the leukaemia immune microenvironment through multiomics (epigenomics transcriptomics, proteomics, metabolomics) and assess its contribution to the effect of the combination of azacitidine and venetoclax.

DETAILED DESCRIPTION:
Study Objective: To decipher the cellular composition of the bone marrow microenvironment before and after treatment with azacitidine and venetoclax. Objective 2: To functionally validate the cellular composition of the bone marrow environment and its contribution in response to treatment using an in vitro model. Objective 3: To evaluate the association between the cellular composition of the bone marrow environment and the achievement of clinical response. Objective 4: To investigate whether the cellular composition of the bone marrow environment and its contribution in response to treatment is associated with lower survival at 18 months. The primary endpoint will be the discovery of the mechanisms of the microenvironment of susceptibility to immunotherapy and their correlation with clinical response (achievement of CR or refractoriness) and survival data. More specifically:

1. Pan-tissue AHR signature - Pan-tissue AHR signature levels will be measured at T1 and T2 using iterative cycles of computational biology analysis and experimental validation. In particular, expression levels will be measured and a cut-off will be set for genes differentially expressed at log2 fold change;
2. The expression level of IFN-y in AML cells (% positive cells) and IDO1 in MSCs (mRNA levels mRNA levels) will be measured at T1 and T2. The expression of IDO1 will be measured in relation to the infiltration of Treg into the bone marrow. A cutoff for IFN-y and IDO1 expression will be set at 30% with fold-change>2 at T2 over T1;
3. The effects of IDO1 inhibitor on metabolic reactivation of effector T cells will be measured at T1 and T2 via mTOR activation. The following parameters will be measured in percentage: 1) glucose dependence, 2) mitochondrial dependence 3) glycolytic capacity and 4) fatty acid and AA oxidation capacity to determine the metabolic state. It will be evaluated the fold change between T2 and T1 of these 4 parameters; STUDY DESIGN This is a prospective, multicentre, tissue-based study aimed at collecting and characterising human tissues isolated from patients with acute myeloid leukaemia, who will receive azacitidine and venetoclax as the standard treatmentv as part of normal clinical practice. Specifically, in addition to the visits as part of normal clinical practice, samples of 80 mL of PB, 45 mL of BM and 1.5 mL of urine in addition to the scheduled blood samples. Samples will be collected at diagnosis (T1) and at the time of treatment response assessment = after the second cycle with azacitidine and venetoclax (T2). Treatment response will be assessed on the basis of the criteria standard response criteria for acute myeloid leukaemia according to the 2022 recommendations of a group of international experts on behalf of European LeukemiaNet25.Patients will be followed up for survival data. The source of survival data will be the patient's medical record. The study will include newly diagnosed, untreated adult patients with acute myeloid leukaemia who are not eligible for chemotherapy, candidates to receive the combination of venetoclax and azacitidine according to standard clinical practice and regardless of study participation. Patients will be enrolled at the time of disease diagnosis. For healthy donors, a total of a total of 60 buffy coats over 24 months. All patients who do not receive treatment (T2) will be excluded from the study. All 60 patients will be considered for the For objectives 2, 3 and 4, only patients who have completed both cycles of therapy will be considered. who have completed both cycles of therapy. The enrolment period of the subjects participating study subjects will be 18 months, the sample collection period will be 2 months, the clinical data analysis period will be 4 months, the clinical data analysis period will be 4 months, the follow-up period will be 12 months, for a total study duration of 36 months.

The study is funded by 'TRANSCAN-3 ERA-NET: supported collaboration of national national and regional programmes in cancer research'; Joint Transnational Call 2021 (JTC 2021) co-funded by the European Commission/DG Research and Innovation: 'Next generation cancer immunotherapy: Targeting the tumour microenvironment'.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age
* Subject has a new diagnosis of AML according to World Health Organization 2022 criteria
* Subject is ineligible for intensive induction chemotherapy according to investigator assessment
* Subject will undergo front-line treatment with azacitidine and venetoclax according to normal clinical practice
* Subject providing signed written informed consent according to ICH/EU/GCP and national local laws

For healthy donors:

* Age ≥ 18 years
* Subject providing signed written informed consent according to ICH/EU/GCP and national local laws

Exclusion Criteria:

For patients:

* Subject has acute promyelocytic leukemia
* Subject has known AML with central nervous system involvement
* Subject has not initiated treatment with azacitidine and venetoclax

For healthy donors:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The planned population size for the study is of 60 prospectively enrolled AML patients. The project outcomes will be evaluated at T2 and correlated with CR and refractoriness obtained at T2 and with survival data obtained at follow-up. Power analysis conducted using Stata 17 indicated that a sample size of n=60 allows at least 0.90 power for the estimation of a linear regression model with 4 to 10 covariates and an expected R2 of 0.30 to 0.75 with α=0.05.
  This linear regression model will include as dependent an immune microenvironment variable measured at T2, and as exposure the treatment variable. By including among covariates the baseline values of the dependent variable we expect to obtain high R2 values
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Pan-tissue AHR signature | At visit 1 (T1, diagnosis), and after the second cycle with azacitidine and venetoclax (T2, 2 months after treatment initiation)
  Pan-tissue AHR signature levels will be measured by using iterative cycles of computational biology analyses and experimental validation (24). In particular, the levels of expression will be detected and a cutoff for differentially expressed genes will be set at log2 fold change.
IFN-y pathway response | At visit 1 (T1), and after the second cycle with azacitidine and venetoclax (T2, 2 months after treatment initiation)
  Expression level of IFN-y in AML cells (% of positive cells) and IDO1 in MSCs (mRNA levels) will be measured. IDO1 expression will be measured in relation to BM Treg infiltration (25).A cutoff for IFN-y and IDO1 expression will be set at 30% with fold-change>2 at T2 over T1.
Immunometabolic shift in T-cells | At visit 1 (T1), and after the second cycle with azacitidine and venetoclax (T2, 2 months after treatment initiation)
  The effects of IDO1 inhibitor for the metabolic re activation of effector T cells will be measured via mTOR activation. We will measure the following parameters as percentages(%): 1) glucose dependence, 2) mitochondrial dependence 3) glycolytic capacity and 4) fatty acid and AA oxidation capacity to determine the metabolic status. The fold change between T2 and T1 of these 4 parameters will be evaluated.
Clinical response | After the second cycle with azacitidine and venetoclax (T2, 2 months after treatement initiation )
  1. Complete Remission (CR): BM blasts <5%; absence of circulating blasts or blasts with Auer rods; absence of extramedullary disease; ANC ≥1.0 x 109
     * L (1,000/μL); platelet count
       ≥100 x 109
     * L (100,000/μL)
  2. CR with partial hematologic recovery (CRh): ANC ≥0.5 x 109
     * L (500/μL) and platelet count ≥50 x 109
     * L (50,000/μL), otherwise all other CR criteria met
  3. CR with incomplete hematologic recovery (CRi): All CR criteria except for residual neutropenia <1.0 x 109
     * L (1,000/μL) or thrombocytopenia <100 x 109
     * L (100,000/μL)
  4. Refractoriness: No CR, CRh or CRi
Survival (Aim 4) | At follow-up (up to 12 months)
  OS (%, months) and RFS (%, months)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Curti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy